CLINICAL TRIAL: NCT04589611
Title: Translating Metabolic Responses to Mechanical Insult Into Early Interventions to Prevent PTOA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: J L Marsh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, J L Marsh, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 201911366
Record Dates: First submitted 2020-06-23; First posted 2020-10-19 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis; Post-traumatic Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Phase I: 6 patients will be treated with single dose open label, and safety measures will be assessed.
  Phase IIa: Once initial safety is confirmed, 20 amobarbital:10 control patients will be treated with the single dose at the initial operation. Patients and attending surgeons will be blinded to the identity of the dose. Assuming continued safety, an additional 20 amobarbital: 10 control patients will be treated with two doses and evaluated. The second dose of 2.5 mM amobarbital will be administered during the second operation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I single amobarbital/Gel-One dose (Experimental): Phase I: An open label study of 3 patients will be done. If no dose limiting toxic (DLT) side effects occur, then an additional 3 patients will be done. If no DLT events occur, the study will proceed to Phase II.
  Interventions: Drug: amobarbital/Gel-One (one dose)
- Phase IIa Part 1 amobarbital/Gel-One dose (Active Comparator): 20 subjects will be randomized to amobarbital/Gel-One single dose.
  Interventions: Drug: amobarbital/Gel-One (one dose)
- Phase IIa Part 1 Placebo (Placebo Comparator): 10 subjects will be randomized to amobarbital/Gel-One single dose.
  Interventions: Drug: Placebo (single dose)
- Phase IIa Part 2 amobarbital/Gel-One dose (Active Comparator): 20 subjects will be randomized to one dose of amobarbital/Gel-One during the initial surgical intervention. A second dose will be administered during the second surgical intervention.
  Interventions: Drug: amobarbital/Gel-One (two doses)
- Phase IIa Part 2 placebo (Placebo Comparator): 20 subjects will be randomized to one dose of placebo during the initial surgical intervention. A second dose will be administered during the second surgical intervention.
  Interventions: Drug: Placebo (two doses)

INTERVENTIONS:
Drug: amobarbital/Gel-One (one dose) — One dose of amobarbital/Gel-One during the initial surgical intervention
  Arms: Phase I single amobarbital/Gel-One dose; Phase IIa Part 1 amobarbital/Gel-One dose
Drug: Placebo (single dose) — One dose of placebo during the initial surgical intervention
  Arms: Phase IIa Part 1 Placebo
Drug: amobarbital/Gel-One (two doses) — One dose of amobarbital/Gel-One during the initial surgical intervention. A second dose will be administered during the second surgical intervention.
  Arms: Phase IIa Part 2 amobarbital/Gel-One dose
Drug: Placebo (two doses) — One dose of placebo during the initial surgical intervention. A second dose will be administered during the second surgical intervention.
  Arms: Phase IIa Part 2 placebo

SUMMARY:
This is a small-scale proof-of concept clinical trial of amobarbital as a treatment to prevent post-traumatic osteoarthritis in fractured ankle joints. The study is a double blind, prospective, randomized, placebo-controlled, stepwise trial. Amobarbital will be delivered to ankle joints in solution with hyaluronic acid (HA) as a vehicle. Amobarbital/HA injections (active dose) will be compared to HA alone (placebo dose). Our primary goal is to confirm safety, but we will also assess whether treatment improves chondrocyte viability and decreases synovial inflammation. The intervention that will be utilized has proven to be effective using vitro and in vivo models. The study team will assess safety and begin to evaluate efficacy of amobarbital/Gel-One in patients having sustained tibial pilon fractures. The study team will use advanced imaging-based methods we have developed to characterize how joints subjected to varying levels of fracture severity and residual elevated contact stress respond in treated and control groups.

DETAILED DESCRIPTION:
This is a small-scale proof-of concept clinical trial of amobarbital as a treatment to prevent post-traumatic osteoarthritis in fractured ankle joints. The study is a double blind, prospective, randomized, placebo-controlled, stepwise trial. Amobarbital will be delivered to ankle joints in solution with hyaluronic acid (HA) as a vehicle. Amobarbital/HA injections (active dose) will be compared to HA alone (placebo dose). Our primary goal is to confirm safety, but we will also assess whether treatment improves chondrocyte viability and decreases synovial inflammation. The intervention that will be utilized has proven to be effective using vitro and in vivo models. The study team will assess safety and begin to evaluate efficacy of amobarbital/Gel-One in patients having sustained tibial pilon fractures. The study team will use advanced imaging-based methods we have developed to characterize how joints subjected to varying levels of fracture severity and residual elevated contact stress respond in treated and control groups.

Phase I:6 subjects will be treated with a single dose open label, and safety measures will be assessed.

Phase II: Once initial safety is confirmed, 20 amobarbital:10 control subjects will be treated with the single dose at the initial operation.

Assuming continued safety, an additional 20 amobarbital:10 control subjects will be treated with two doses and evaluated. The second dose of 2.5 mM amobarbital will be administered during the second operation.

Subjects will participate in the following procedures:

SOC surgical intervention Randomization to Amobarbital/Gel-One arm or control arm X-rays CT scans Blood and urine Questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Acute closed or type 1 open ankle fractures (classified as OTA/AO 43 B 1-3 and 43 C 1- 3 or classified as 42 B and C fractures with 25% talar displacement and one of the following; syndesmosis injury or medial malleolar fracture at or above the shoulder) (Marsh et al., 2007)) without operative ipsilateral extremity trauma
* Posterior malleolar and supination adduction rotational fractures that have an articular fracture line across the articular surface of the distal tibia. Posterior malleolar fractures should affect 25% of the articular surface or greater.
* Fractures must have initial treatment within 72 hours of injury including initial injection of amobarbital or placebo.

Exclusion Criteria:

* Diabetes
* Pregnant or nursing mothers and individuals with child-bearing potential that are not using birth control methods with >99% efficacy.
* Allergy to poultry products or cinnamon
* Previous injuries to the ankle
* High grade open wounds
* Pre-existing immunologic or hematologic diseases
* Pre-existing ankle arthritis
* Ipsilateral fractures
* Associated injuries that preclude standard rehabilitation
* Pre-existing dysfunction of the kidneys, liver, blood, immune system, endocrine system (excluding diabetes)
* Serum creatinine >/= 1.4 mg/dl; BUN > 30 mg/dl; ALT >/= 60 IU/L in males and >/= 50 IU/L in females; AST >/= 45 IU/L in males and > 40 IU/L in females; bilirubin > 1.3 mg/dL; platelets </= 50,000/ul; glucose > 200 mg/dL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Determine the number of participants with systemic adverse events including the change in laboratory values to assess the systemic safety of amobarbital. | Pre-op baseline on the day before external fixation surgery (within 24 hours of injury), immediately post-op, and at 1, 2, and 4 days post-op. At the time of internal fixation (3-21 days after external fixation) and at 1, 2, and 4 days post-op.]
  By using CBC and standard clinical chemistry assays to quantify circulating, ALT, AST, Bilirubin, Creatinine, and BUN and the measurement of urine protein content, the number of participants that have abnormal laboratory values will be determined.
Determine the number of participants with a change of local toxicity in tissues. | Pre-op baseline on the day before external fixation surgery (within 24 hours of injury), immediately post-op, and at 1, 2, and 4 days post-op. At the time of internal fixation (3-21 days after external fixation) and at 1, 2, and 4 days post-op.
  By using osteochondral fragments obtained during the internal fixation surgery, local toxicity will be determined by examining the tissue for cartilage and synovial histological changes.

SECONDARY OUTCOMES:
Patient Reported Outcome Measurement Information Systems (PROMIS) - Pain Interference | 3, 6, 12, and 24 months
  Description: Pain interference 6 questions 5 pt scale - the higher the score the greater the pain
Patient Reported Outcome Measurement Information Systems (PROMIS) Physical Function | Global Health - T-score - mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. Higher is better.
  Physical Function - T-score - mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. Higher is better.
Patient Reported Outcome Measurement Information Systems (PROMIS) Global Health questionnaires. | 3, 6, 12, and 24 months
  Global Health - T-score - mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. Higher is better.
American Orthopaedic Foot and Ankle Society (AOFAS) Score. | 3, 6, 12, and 24 months
  0-100 point scale with 100 perfect ankle function
Foot and Ankle Disability Index (FADI). | 3, 6, 12, and 24 months
  Description: total 104 points scored in a percentage scale with 100% perfect
X-Ray based Kellgren-Lawrence Grade | 3, 6, 12, and 24 months
  Radiograph imaging graded on scale 1 (no arthritis)-4 (severe arthritis)
CT-based fracture energy | 6 months
  Fracture energy is measured in Joules. It is from CT data and measured computationally. It is a continuous measure - Higher Joules = more energy = worse fracture
CT-based Contact Stress | 6 months
  Vertical CT scan of ankle are segmented and analyzed using finite element analysis. Results are expressed as Contract Stress Exposure (MPa) across areas.
CT-based Joint Space Width | 6 months
  Vertical CT scan of ankle used to measure Joint Space Width at several locations to measure distance to calculate the mean tibiotalar joint space (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified radiographic and clinical data will be shared.